CLINICAL TRIAL: NCT02288949
Title: STratification AND Outcome of Patients With the Acute Respiratory Distress Syndrome
Brief Title: Stratification of the Acute Respiratory Distress Syndrome
Acronym: STANDARDS
Status: Completed | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Collaborators: Asociación Científica Pulmón y Ventilación Mecánica (Other)
Responsible Party: Principal Investigator, Jesus Villar, Director, Multidisciplinary Organ Dysfunction Evaluation Research Network, Dr. Negrin University Hospital
Other Study IDs: ACPVM-2014
Record Dates: First submitted 2014-11-05; First posted 2014-11-13 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: mechanical ventilation, stratificacion, lung severity
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Vernalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prospective cohort: Stratification of patients admitted into a network of Spanish ICUs.
  Interventions: Other: stratification

INTERVENTIONS:
Other: stratification — Patients will be stratified based on the values of relevant demographics, pulmonary and systemic variables in relation to mortality in the intensive care unit.

SUMMARY:
The American-European Consensus Conference (AECC) and the Berlin definitions of the Acute Respiratory Distress Syndrome (ARDS) could be adequate for epidemiologic studies, but it is not adequate for inclusion of patients into therapeutic clinical trials. Despite recent reports on the effects of standardized ventilator settings on PaO2/FIO2 and fulfillment of AECC and Berlin definitions of ARDS, it is still a matter of debate whether the assessment of hypoxemia at 24 hours is the most appropriate tool for stratifying lung severity in patients with ARDS. The investigators will perform an observational, multicenter, prospective audit in a network of intensive care units in Spain and China for validating and confirming that the assessment of hypoxemia at 24 hours after ARDS onset is the most valuable tool for stratifying and predicting outcome in patients with ARDS.

DETAILED DESCRIPTION:
In 1994, the American-European Consensus Conference (AECC) defined ARDS as follows: 1) acute and sudden onset of severe respiratory distress, 2) bilateral infiltrates on frontal chest radiograph, 3) absence of left atrial hypertension or no clinical signs of left heart failure, and 4) severe hypoxemia, as PaO2/FiO2 ratio <200 mmHg, regardless of FIO2 or PEEP levels. Although this definition could be adequate for epidemiologic studies, it is not adequate for inclusion of patients into therapeutic clinical trials. In 2012, a proposal for updating the ARDS definition (the Berlin criteria) was published and an empirical classification was proposed according to three PaO2/FiO2 cut-off values at ARDS onset: severe (≤100 mmHg), moderate (>100-≤200), and mild (>200-≤300) on PEEP≥5 cmH2O. However, despite that there is sufficient evidence about the interactions between PEEP and FiO2, the Berlin criteria did not mandate the assessment of hypoxemia at 24 hours under standarized guidelines.

The PaO2/FIO2 can be easily manipulated. Alterations in PEEP and FIO2 can dramatically change the PaO2/FIO2. Despite recent reports on the effects of standardized ventilator settings on PaO2/FIO2 and fulfillment of AECC definitions of ARDS, it is still a matter of debate whether the assessment of hypoxemia at 24 hours is the most appropriate tool for stratifying lung severity in patients with ARDS.

The investigators will examine whether the assessment of hypoxemia at 24 h after ARDS diagnosis under standard guidelines for ventilatory management have an impact on the stratification of lung severity and on predicting mortality of ARDS patients in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the AECC definition for ARDS on PEEP greater or equal than 5 cmH2O (or the Berlin criteria for moderate and severe ARDS).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive ARDS patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
range of values of variables associated with the highest or lowest mortality | within the first 24 h of ARDS onset

SECONDARY OUTCOMES:
stratification by risk of death based on variables associated with worst outcome | ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Villar, MD, PhD, Principal Investigator — Hospital Universitario Dr. Negrin
Locations (1):
- Hospital Virgen de la Luz, Cuenca, Spain

REFERENCES:
- [Derived] Villar J, Gonzalez-Martin JM, Ambros A, Mosteiro F, Martinez D, Fernandez L, Soler JA, Parra L, Solano R, Soro M, Del Campo R, Gonzalez-Luengo RI, Civantos B, Montiel R, Pita-Garcia L, Vidal A, Anon JM, Ferrando C, Diaz-Dominguez FJ, Mora-Ordonez JM, Fernandez MM, Fernandez C, Fernandez RL, Rodriguez-Suarez P, Steyerberg EW, Kacmarek RM; Spanish Initiative for Epidemiology, Stratification and Therapies of ARDS (SIESTA) Network. Stratification for Identification of Prognostic Categories In the Acute RESpiratory Distress Syndrome (SPIRES) Score. Crit Care Med. 2021 Oct 1;49(10):e920-e930. doi: 10.1097/CCM.0000000000005142. PMID 34259448
- [Derived] Villar J, Ambros A, Mosteiro F, Martinez D, Fernandez L, Ferrando C, Carriedo D, Soler JA, Parrilla D, Hernandez M, Andaluz-Ojeda D, Anon JM, Vidal A, Gonzalez-Higueras E, Martin-Rodriguez C, Diaz-Lamas AM, Blanco J, Belda J, Diaz-Dominguez FJ, Rico-Feijoo J, Martin-Delgado C, Romera MA, Gonzalez-Martin JM, Fernandez RL, Kacmarek RM; Spanish Initiative for Epidemiology, Stratification and Therapies of ARDS (SIESTA) Network. A Prognostic Enrichment Strategy for Selection of Patients With Acute Respiratory Distress Syndrome in Clinical Trials. Crit Care Med. 2019 Mar;47(3):377-385. doi: 10.1097/CCM.0000000000003624. PMID 30624279
- [Derived] Villar J, Martinez D, Mosteiro F, Ambros A, Anon JM, Ferrando C, Soler JA, Montiel R, Vidal A, Conesa-Cayuela LA, Blanco J, Arrojo R, Solano R, Capilla L, Del Campo R, Civantos B, Fernandez MM, Aldecoa C, Parra L, Gutierrez A, Martinez-Jimenez C, Gonzalez-Martin JM, Fernandez RL, Kacmarek RM; Stratification and Outcome of Acute Respiratory Distress Syndrome (STANDARDS) Network. Is Overall Mortality the Right Composite Endpoint in Clinical Trials of Acute Respiratory Distress Syndrome? Crit Care Med. 2018 Jun;46(6):892-899. doi: 10.1097/CCM.0000000000003022. PMID 29420341